CLINICAL TRIAL: NCT03245398
Title: Efficacy and Safety of a Single-dose Regimen and a Multi-dose Regimen of Mebendazole Against Hookworm Infections in School Children: a Randomized Controlled Trial
Brief Title: Efficacy and Safety of a Multi-dose Regimen of Mebendazole Against Hookworm in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jennifer Keiser (Other)
Collaborators: PATH (Other); Public Health Laboratory Ivo de Carneri (Other)
Responsible Party: Sponsor-Investigator, Jennifer Keiser, Dr., Swiss Tropical & Public Health Institute
Organization: Swiss Tropical & Public Health Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRIPLEMEB_PEMBA
Record Dates: First submitted 2017-07-22; First posted 2017-08-10 (Actual); Results first posted 2019-06-17 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-03

CONDITIONS: Hookworm
MeSH Terms: conditions — Ancylostomiasis | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, physicians, nurses and investigators will all be blinded. Based on the randomization list, individual envelopes with the correct combination of mebendazole tablets and placebos will be prepared. The randomization code is then sealed in an envelope. Unblinding will only occur in case of a SAE, SUSAR or other kind of emergency.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single dose of mebendazole (Active Comparator): In day 1 each child in this treatment arm will receive a 500 mg tablet of mebendazole plus one 100 mg placebo tablet in the morning. In the afternoon of day 1 they will only receive the placebo. In day 2 and 3 each child will receive one placebo twice a day (in the morning and in the evening)
  Interventions: Drug: Treatment with one of the two regimens of mebendazole
- Multiple dose of mebendazole (Active Comparator): In day 1 each child in this treatment arm will receive a 100 mg tablet of mebendazole plus one 500 mg placebo tablet in the morning. In the afternoon of day 1 they will only receive the 100 mg tablet of mebendazole. In day 2 and 3 each child will receive one 100 mg tablet of mebendazole twice a day (in the morning and in the evening).
  Interventions: Drug: Treatment with one of the two regimens of mebendazole

INTERVENTIONS:
Drug: Treatment with one of the two regimens of mebendazole — Once in the morning and once in the evening for 3 consecutive days

SUMMARY:
This study is a double-blind randomized clinical trial which aims at providing evidence on the efficacy and safety of two regimens of mebendazole in school-aged children. Thus, our primary objective is to assess the efficacy and safety of: i) 100 mg solid tablets twice a day for 3 days, and ii) one dose of 500 mg solid tablets of mebendazole in participants aged 6-12, inclusive, infected with hookworm.

The primary endpoint of the trial is the cure rate (CR) of the 3-day regimen of mebendazole against hookworm and a single dose mebendazole treatment.

The secondary objectives are to determine if the multi-dose regimen is superior to the single dose regimen, evaluate the efficacy against concomitant soil-transmitted helminth infections, and assess the safety of both mebendazole regimens.

After obtaining informed consent from children's caregiver, the medical history of the participating individuals will be assessed with a standardized questionnaire, in addition to a clinical examination carried out by the study physician on the treatment day. Enrollment will be based on two stool samples which will be collected, if possible, on two consecutive days or otherwise within a maximum of 5 days apart. All stool samples will be examined with duplicated Kato-Katz thick smears by experienced laboratory technicians.

Randomization of participants into the two treatment arms will be stratified according to intensity of infection. Participants will be interviewed before treatment for clinical symptoms and 3 hours after every morning treatment and 24 hours after every morning treatment about the occurrence of adverse events. The efficacy of the treatment will be determined 14-21 days post-treatment by collecting another two stool samples.

The primary analysis will include all participants with primary end point data (available case analysis). Supplementary, two sensitivity analyses will be conducted imputing all missing endpoint data as treatment failures or all as treatment success. CRs will be calculated as the percentage of egg-positive participants at baseline who become egg-negative after treatment. CRs will be compared by using unadjusted logistic regression. To assess model robustness with respect to covariates, adjusted logistic regressions (adjustment for age, sex, school, weight and strata) will be performed.

Geometric and arithmetic mean egg counts will be calculated for the different treatment arms before and after treatment to assess the corresponding ERRs. Bootstrap resampling method with 5,000 replicates will be used to calculate 95% confidence intervals (CIs) for ERRs and the difference of the ERRs.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent signed by parents and/or caregiver; and oral assent by participant.
* Able and willing to be examined by a study physician at the beginning of the study.
* Able and willing to provide two stool samples at the beginning (baseline) and approximately three weeks after treatment (follow-up).
* Positive for hookworm eggs in the stool (≥ 100 EPG and at least two Kato-Katz thick smears slides with more than one hookworm egg).
* Absence of major systemic illnesses, e.g. diabetes, severe anemia (HB<8.0 g/l) as assessed by a medical doctor at school, upon initial clinical assessment.
* No known or reported history of chronical illness as cancer, diabetes, chronic heart, liver or renal disease.
* No recent anthelminthic treatment (within past 4 weeks). No known allergy to study medications (mebendazole and albendazole).

Exclusion Criteria:

No written informed consent by parents and/or caregiver; no oral assent by participant.

* Menarche, based on self-report
* Presence of major systemic illnesses, e.g. diabetes, severe anemia (HB<8.0 g/l) as assessed by a medical doctor, upon initial clinical assessment.
* History of acute or severe chronic disease.
* Recent use of anthelminthic drug (within past 4 weeks).
* Attending other clinical trials during the study.
* Negative diagnostic result for hookworm eggs in the stool (< 100 EPG (total of the four slides) and/or only one Kato-Katz thick smear slide with more than one hookworm egg).

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 186 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2017-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Keiser, PhD, Principal Investigator — Swiss Tropical & Public Health Institute
Locations (1):
- Public Health Laboratory Ivo de Carneri, P.O. Box 122, Chake Chake, Pemba, Tanzania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Palmeirim MS, Ame SM, Ali SM, Hattendorf J, Keiser J. Efficacy and Safety of a Single Dose versus a Multiple Dose Regimen of Mebendazole against Hookworm Infections in Children: A Randomised, Double-blind Trial. EClinicalMedicine. 2018 Jul 11;1:7-13. doi: 10.1016/j.eclinm.2018.06.004. eCollection 2018 Jul. PMID 31193620

RESULTS

PARTICIPANT FLOW:
Groups:
- Single 500 mg Dose of Mebendazole: In the morning of day 1 each child in this treatment arm received a 500 mg tablet of mebendazole plus one 100 mg placebo tablet. In the afternoon of day 1 they only received the placebo. In day 2 and 3 each child received one placebo tablet twice a day (in the morning and in the evening).
  Treatment with one of the two regimens of mebendazole: Once in the morning and once in the evening for 3 consecutive days
- Multiple (Bid for 3 Days) Dose of 100 mg Mebendazole: In the morning of day 1 each child in this treatment arm received a 100 mg tablet of mebendazole plus one 500 mg placebo tablet. In the afternoon of day 1 they only received the 100 mg tablet of mebendazole. In day 2 and 3 each child received one 100 mg tablet of mebendazole twice a day (in the morning and in the evening).
  Treatment with one of the two regimens of mebendazole: Once in the morning and once in the evening for 3 consecutive days
Period: Overall Study
Arm/Group | Single 500 mg Dose of Mebendazole | Multiple (Bid for 3 Days) Dose of 100 mg Mebendazole
Started | 93 | 93
Completed | 92 | 93
Not Completed | 1 | 0
Not completed — Travelled to another island | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single 500 mg Dose of Mebendazole | Multiple (Bid for 3 Days) Dose of 100 mg Mebendazole | Total
Number analyzed (Participants) | 93 | 93 | 186
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.1 (1.6) | 10.1 (1.6) | 10.1 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 46 | 85
  Male | 54 | 47 | 101
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 93 | 93 | 186
Region of Enrollment [Number; unit: participants]
  Tanzania | 93 | 93 | 186
Mean weight (kg) [Mean (Standard Deviation); unit: kg] | 26.7 (5.3) | 26.2 (5.1) | 26.4 (5.2)
Mean height (cm) [Mean (Standard Deviation); unit: cm] | 132.0 (10.2) | 131.8 (9.6) | 131.9 (9.9)
Infected with hookworm [Count of Participants; unit: Participants] | 93 | 93 | 186
Median EPG hookworm [Median (Inter-Quartile Range); unit: Eggs per gram (EPG)] | 222 [78 to 534] | 222 [96 to 606] | 222 [90 to 582]
EPG hookworm (geometric mean) [Geometric Mean (Full Range); unit: EPG] | 219 [172 to 279] | 234 [185 to 297] | 226 [191 to 268]
Light hookworm infection (1-1999 EPG) [Count of Participants; unit: Participants] | 89 | 90 | 179
Moderate hookworm infection (2000-3999 EPG) [Count of Participants; unit: Participants] | 3 | 3 | 6
Heavy hookworm infection (≥4000 EPG) [Count of Participants; unit: Participants] | 1 | 0 | 1
Infected with T. trichiura [Count of Participants; unit: Participants] | 88 | 91 | 179
EPG T. trichiura (geometric mean) [Geometric Mean (Full Range); unit: EPG] | 661.8 [541 to 809] | 725.7 [574 to 918] | 693 [595 to 808]
Light T. trichiura infection (1-999 EPG) [Count of Participants; unit: Participants] | 59 | 56 | 115
Moderate T. trichiura infection (1000-9999 EPG) [Count of Participants; unit: Participants] | 30 | 35 | 65
Heavy T. trichiura infection (≥10,000 EPG) [Count of Participants; unit: Participants] | 0 | 0 | 0
Infected with A. lumbricoides [Count of Participants; unit: Participants] | 47 | 51 | 98
EPG A. lumbricoides (geometric mean) [Geometric Mean (Full Range); unit: EPG] | 2691.2 [1379 to 5251] | 4095.9 [2233 to 7513] | 3349 [2148 to 5219]
Light A. lumbricoides infection (1-4999 EPG) [Count of Participants; unit: Participants] | 28 | 20 | 48
Moderate A. lumbricoides infection (5000-49,999 EPG) [Count of Participants; unit: Participants] | 15 | 28 | 43
Heavy A. lumbricoides infection (≥50,000 EPG) [Count of Participants; unit: Participants] | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Cure Rate (CR) of Mebendazole Against Hookworm
Description: Cure rates (CRs) will be calculated as the percentage of egg-positive participants at baseline who become egg-negative after treatment.
Time Frame: baseline (before treatment) and 18 to 22 days post-treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants cured
Arm/Group | Single 500 mg Dose of Mebendazole | Multiple (Bid for 3 Days) Dose of 100 mg Mebendazole
Number analyzed (Participants) | 92 | 93
percentage of participants cured | 13 [6.9 to 21.7] | 97.9 [92.4 to 99.7]

2. Secondary Outcome: Geometric Mean Egg Reduction Rate (ERR) of the Two Regimens of Mebendazole Against Hookworm
Description: Eggs per gram of stool (EPG) will be assessed by adding up the egg counts from the quadruplicate Kato-Katz thick smears and multiplying this number by a factor of six. The egg reduction rate (ERR) is calculated as follows: ERR = (1-(geometric mean EPG at follow-up/geometric mean EPG at baseline))*100). Note: in contrast to the publication the "outcome measure" entry mask requires the complementary percentage: (geometric mean at follow-up/geometric mean at baseline)*100).
Time Frame: baseline (before treatment) and 18 to 22 days post-treatment
Measure: Geometric Mean (95% Confidence Interval); unit: percentage change
Arm/Group | Single 500 mg Dose of Mebendazole | Multiple (Bid for 3 Days) Dose of 100 mg Mebendazole
Number analyzed (Participants) | 92 | 93
percentage change | -68.0 [-78.6 to -51.5] | -100 [-100 to -99.9]

3. Secondary Outcome: CR of Both Mebendazole Regimens Against Trichuris Trichiura
Description: as for outcome 1
Time Frame: baseline (before treatment) and 18 to 22 days post-treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants cured
Arm/Group | Single 500 mg Dose of Mebendazole | Multiple (Bid for 3 Days) Dose of 100 mg Mebendazole
Number analyzed (Participants) | 92 | 93
percentage of participants cured | 6.8 [4.6 to 17.8] | 42.9 [33.8 to 54.8]

4. Secondary Outcome: Geometric ERR of Both Mebendazole Regimens Against Trichuris Trichiura
Description: as for outcome 2
Time Frame: baseline (before treatment) and 18 to 22 days post-treatment
Measure: Mean (95% Confidence Interval); unit: percentage of change
Arm/Group | Single 500 mg Dose of Mebendazole | Multiple (Bid for 3 Days) Dose of 100 mg Mebendazole
Number analyzed (Participants) | 92 | 93
percentage of change | -71.7 [-78.5 to -56.7] | -98.1 [-98.7 to -96.8]

5. Secondary Outcome: Cure Rate (CR) of Both Mebendazole Regimens Against Ascaris Lumbricoides
Description: as for outcome 1
Time Frame: baseline (before treatment) and 18 to 22 days post-treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants cured
Arm/Group | Single 500 mg Dose of Mebendazole | Multiple (Bid for 3 Days) Dose of 100 mg Mebendazole
Number analyzed (Participants) | 92 | 93
percentage of participants cured | 100 [100 to 100] | 98 [94.2 to 100]

6. Secondary Outcome: Geometric ERR of Both Mebendazole Regimens Against Ascaris Lumbricoides.
Description: as for outcome 2
Time Frame: baseline (before treatment) and 18 to 22 days post-treatment
Measure: Mean (95% Confidence Interval); unit: percentage change
Arm/Group | Single 500 mg Dose of Mebendazole | Multiple (Bid for 3 Days) Dose of 100 mg Mebendazole
Number analyzed (Participants) | 92 | 93
percentage change | -100 [-100 to -100] | -100 [-100 to -100]

7. Secondary Outcome: Arithmetic ERR of the Two Regimens of Mebendazole Against Hookworm
Description: Eggs per gram of stool (EPG) will be assessed by adding up the egg counts from the quadruplicate Kato-Katz thick smears and multiplying this number by a factor of six. The egg reduction rate (ERR) is calculated as follows: ERR = (1-(arithmetic mean EPG at follow-up/arithmetic mean EPG at baseline))*100). Note: in contrast to the publication the "outcome measure" entry mask requires the complementary percentage: (arithmetic mean at follow-up/arithmetic mean at baseline)*100).
Time Frame: baseline (before treatment) and 18 to 22 days post-treatment
Measure: Mean (95% Confidence Interval); unit: percentage change
Arm/Group | Single Dose of Mebendazole | Multiple Dose of Mebendazole
Number analyzed (Participants) | 92 | 93
percentage change | -52.7 [-63.6 to -40.3] | -99.8 [-100 to -99.3]

8. Secondary Outcome: Arithmetic ERR of Both Mebendazole Regimens Against Trichuris Trichiura
Description: as for outcome 7
Time Frame: baseline (before treatment) and 18 to 22 days post-treatment
Measure: Mean (95% Confidence Interval); unit: percentage change
Arm/Group | Single 500 mg Dose of Mebendazole | Multiple (Bid for 3 Days) Dose of 100 mg Mebendazole
Number analyzed (Participants) | 92 | 93
percentage change | -49.1 [-61.0 to -31.7] | -91.6 [-94.6 to -88.4]

9. Secondary Outcome: Arithmetic ERR of Both Mebendazole Regimens Against Ascaris Lumbricoides
Description: as for outcome 7
Time Frame: baseline (before treatment) and 18 to 22 days post-treatment
Measure: Mean (95% Confidence Interval); unit: percentage change
Arm/Group | Single 500 mg Dose of Mebendazole | Multiple (Bid for 3 Days) Dose of 100 mg Mebendazole
Number analyzed (Participants) | 92 | 93
percentage change | -100 [-100 to -100] | -99.1 [-100 to -96.9]

10. Other Pre Specified Outcome: Comparison of the Sensitivity of Kato Katz to Quantitative Polymerase Chain Reaction (PCR) Assays
Description: Two aliquots (about 1 g of stool each) of positive samples will be stored in ethanol and transported to the Swiss Tropical Public Health Institute for subsequent DNA extraction and diagnostic.
Time Frame: 1 year
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Prevalence of Genetic Resistance Markers Among Participants
Description: The same two aliquots of stool will be used in this section.. Additionally, a Harada Mori culture will be prepared from one of the stool samples of each child at baseline and at follow-up to extract hatched larvae. Larvae will be stored in ethanol. Both stool and larvae samples will undergo an assessment of drug resistance-associated single-nucleotide polymorphisms.
Time Frame: 2 years
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Distribution of Hookworm Species Among Participants
Description: Genetic differentiation between Necator americanus and Ancylostoma duodenale using PCRs will allow us to identify which of the species is most prevalent.
Time Frame: 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data collected 3h after the first treatment time point
Arm/Group | Single 500 mg Dose of Mebendazole | Multiple (Bid for 3 Days) Dose of 100 mg Mebendazole
All-Cause Mortality (participants affected / at risk) | 0/93 | 0/93
Serious Adverse Events (participants affected / at risk) | 0/93 | 0/93
Other Adverse Events (participants affected / at risk) | 2/93 | 8/93
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single 500 mg Dose of Mebendazole (N=93) | Multiple (Bid for 3 Days) Dose of 100 mg Mebendazole (N=93)
Abdominal pain (Gastrointestinal disorders) | 2 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-07-17): https://cdn.clinicaltrials.gov/large-docs/98/NCT03245398/Prot_SAP_ICF_000.pdf